CLINICAL TRIAL: NCT00802204
Title: Dopamine Receptor Availability and Insulin Resistance
Brief Title: Dopamine and Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Julia P.Dunn,MD, Physician, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: IRB#080861 and 061246
Record Dates: First submitted 2008-12-02; First posted 2008-12-04 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-03

CONDITIONS: Obesity
Keywords: Obesity; Insulin Resistance; Neuroendocrine regulation; Eating behaviors; Dopamine signaling
MeSH Terms: conditions — Obesity; Insulin Resistance; Feeding Behavior | interventions — Magnetic Resonance Spectroscopy; Glucose Tolerance Test; Quality of Life; Caloric Restriction

STUDY DESIGN:
Intervention Model Description: Lean who are age and sex similar to obese will complete baseline outcome measurements only.
  Obese will complete baseline outcome measurements then the VLCD intervention with post outcome measurements .
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lean controls (Active Comparator): Lean complete baseline outcome measures only
  Interventions: Radiation: PET scan; Procedure: Oral glucose tolerance test; Procedure: MRI; Behavioral: Psychological scales to assess attitudes and behaviors related to eating and quality of life
- Obese (Experimental): Obese completing baseline and post-VLCD outcome measures
  Interventions: Radiation: PET scan; Procedure: Oral glucose tolerance test; Procedure: MRI; Behavioral: Psychological scales to assess attitudes and behaviors related to eating and quality of life; Other: Caloric Restriction

INTERVENTIONS:
Radiation: PET scan — Both lean and obese undergo a PET scan of the brain using the radioligand,fallypride [18F] at baseline. Obese subjects who complete caloric restriction will have repeat scan after diet.
  Completed at baseline and post-VLCD
Procedure: Oral glucose tolerance test — Subjects will be required to drink a glucose solution; blood samples will be taken over a 5-hour time period Completed at baseline by both lean and obese and in obese post-VLCD
Procedure: MRI — An MRI of the brain and abdomen will be performed prior to PET scan One time at baseline in both lean and obese
Behavioral: Psychological scales to assess attitudes and behaviors related to eating and quality of life — A series of short psychological scales will be administered during the study. Completed at baseline
Other: Caloric Restriction — Obese participants only complete a short-term (~10days) very low calorie diet
  Arms: Obese

SUMMARY:
Obese individuals have fewer striatal dopamine type 2 receptors (DRD2) than normal weight individuals. Lower DRD2 levels are associated with addiction and a decreased sense of pleasure.Obesity is also associated with insulin resistance (poor insulin action).We propose that insulin resistance and low DRD2 are associated. Using PET imaging,we aim to determine DRD2 binding potential (BP) in the brain is associated with insulin resistance and neuroendocrine hormone levels. Obese participants will be compared to lean, gender and age similar participants. We also aim to determine the effect of caloric restriction on DRD2 BP in obese subjects

DETAILED DESCRIPTION:
In has been reported obese individuals have fewer striatal dopamine type 2 receptors (DRD2) compared to normal weight individuals congruent with diet induced obese rodent models and similar to models of addiction. Lower DRD2 levels are associated with addiction and a decreased sense of pleasure. Excessive weight gain also contributes to the onset of impaired insulin signaling (insulin resistance). In the brain insulin regulates monoamines and has trophic effects. We propose that the previous reports of low DRD2 in individuals with obesity will be associated with the degree of insulin resistance. Using PET imaging, we aim to determine DRD2 binding potential (BP) in the striatum and hypothesize these measurements will be associated with insulin resistance and potentially other neuroendocrine hormone levels. Obese participants will be compared to lean, sex and age similar participants. We also aim to determine the effect of caloric restriction on DRD2 BP in obese subjects. We hypothesize the caloric restriction will improve insulin resistance and that changes in DRD2 binding will be associated with changes in insulin signaling.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-60 yrs
* obese BMI > 30kg/m2 and Weight less than 350 lbs
* lean control BMI 18-25kg/m2

Exclusion Criteria:

* Structured exercise > equivalent to 30mins 5x week of walking times a week
* History of Substance Abuse, including but exclusive to alcohol, cocaine, marijuana, heroin, nicotine
* Current psychiatric disorder or significant h/o disorder
* Use or any antidepressants or antipsychotics for last 3-6months or depot antipsychotics in the last 12 months
* Any condition felt by PI or co-investigators to interfere with ability to complete the study
* Inability to abstain from alcohol, physical exercise or > 1 cup of coffee or equivalent daily for 3 days prior to imaging studies
* Significant co-morbidities including atherosclerotic disease, metabolic disease, liver or renal insufficiency or abnormality found on MRI
* Any condition which would interfere with MRI or PET studies, e.g. claustrophobia, cochlear implant, metal fragments in eyes, cardiac pacemaker, neural stimulator, tattoos with iron pigment and metallic body inclusions or other metal implanted in the body which may interfere with MRI scanning
* Subjects on medications determined by PI, ex. sibutramine, frequent benzodiazepines or related drugs, which could affect quality of study for last 3 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-12; Primary Completion 2011-04 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia P Dunn, MD, Principal Investigator — Vanderbilt University Medical Center; Robert M Kessler, MD, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Dunn JP, Abumrad NN, Patterson BW, Kessler RM, Tamboli RA. Brief communication: beta-cell function influences dopamine receptor availability. PLoS One. 2019 Mar 8;14(3):e0212738. doi: 10.1371/journal.pone.0212738. eCollection 2019. PMID 30849082
- [Derived] Dunn JP, Abumrad NN, Kessler RM, Patterson BW, Li R, Marks-Shulman P, Tamboli RA. Caloric Restriction-Induced Decreases in Dopamine Receptor Availability are Associated with Leptin Concentration. Obesity (Silver Spring). 2017 Nov;25(11):1910-1915. doi: 10.1002/oby.22023. Epub 2017 Sep 25. PMID 28944597
- [Derived] Garcia AE, Kasim N, Tamboli RA, Gonzalez RS, Antoun J, Eckert EA, Marks-Shulman PA, Dunn J, Wattacheril J, Wallen T, Abumrad NN, Flynn CR. Lipoprotein Profiles in Class III Obese Caucasian and African American Women with Nonalcoholic Fatty Liver Disease. PLoS One. 2015 Nov 23;10(11):e0142676. doi: 10.1371/journal.pone.0142676. eCollection 2015. PMID 26599819
- [Derived] Dunn JP, Kessler RM, Feurer ID, Volkow ND, Patterson BW, Ansari MS, Li R, Marks-Shulman P, Abumrad NN. Relationship of dopamine type 2 receptor binding potential with fasting neuroendocrine hormones and insulin sensitivity in human obesity. Diabetes Care. 2012 May;35(5):1105-11. doi: 10.2337/dc11-2250. Epub 2012 Mar 19. PMID 22432117

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 lean enroll but only 8 complete. The lean complete study after baseline outcome measurements.
  19 obese enroll but only 18 complete baseline outcome measurements and of these 15 completed the VLCD and post-outcome measurements
Groups:
- Lean: BMI<~25kg/m2
- Obese: BMI>/=30kg/m2
Period: Overall Study
Arm/Group | Lean | Obese
Started | 9 | 19
Completed | 8 | 18
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lean | Obese | Total
Number analyzed (Participants) | 8 | 18 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (9) | 39 (8) | 39 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 18 | 26
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  African American Participants | 1 | 7 | 8
  Caucasian Participants | 7 | 11 | 18
Region of Enrollment [Number; unit: participants]
  United States | 8 | 18 | 26
Weight [Mean (Standard Deviation); unit: kg] | 60 (7) | 104 (17) | 91 (26)
BMI [Mean (Standard Deviation); unit: kg/m2] | 23 (2) | 39 (6) | 33 (9)
Beck Depression Inventory II(BDI-II) [Mean (Standard Deviation); unit: scores on a scale] — 0-63 with higher scores indicating increased depressive symptoms. Scores above 20 indicate moderate depressive symptoms.
  scores on a scale | 3 (5) | 7 (6) | 6 (6)
OGTT_SI (Insulin Sensitivity from OGTT) [Mean (Standard Deviation); unit: (10-4min-1/µU*mL)] — Insulin Sensitivity from Oral Glucose Tolerance Test was estimated using the oral minimal model method
  (10-4min-1/µU*mL) | 11.2 (4.1) | 3.98 (2.7) | 6 (5)
Insulin [Mean (Standard Deviation); unit: (µU/ml)] | 6 (2) | 18 (9) | 14 (10)
Glucose [Mean (Standard Deviation); unit: mg/dl] | 82 (6) | 87 (9) | 86 (8)
Leptin [Mean (Standard Deviation); unit: ng/ml] | 13 (5) | 43 (12) | 34 (18)
Acyl Ghrelin [Mean (Standard Deviation); unit: pg/ml] | 235 (104) | 78 (55) | 132 (106)

OUTCOME MEASURES:

1. Primary Outcome: Striatal DRD2 Receptor Binding
Description: Region of interest compared to reference region to calculate binding potential
Time Frame: Baseline and after 8-10days VLCD
Population: Baseline outcome measurements are compared between lean and obese. Baseline and post outcome measurements are compared for the obese who completed VLCD
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Lean Baseline | Obese Baseline | Obese Post-diet
Number analyzed (Participants) | 8 | 18 | 15
ratio
  caudate | 28 (3) | 33 (3) | 32 (3)
  putamen | 33 (3) | 38 (3) | 36 (4)
  ventral striatum | 19 (4) | 22 (3) | 22 (3)
Statistical Analysis 1: Comparison: Obese Baseline vs Obese Post-diet; Baseline outcome measurements are compared between lean and obese. Baseline and post outcome measurements are compared for the obese who completed VLCD; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; describe
Statistical Analysis 2: Comparison: Obese Baseline vs Obese Post-diet; Paired t-test to compare baseline and post-diet outcome measures; Test type: Other; p < 0.05, t-test, 2 sided

2. Primary Outcome: Insulin
Description: microU/ml
Time Frame: Baseline to post 8-10days after VLCD
Measure: Mean (Standard Deviation); unit: microU/ml
Arm/Group | Lean Baseline | Obese Baseline | Obese Post-diet
Number analyzed (Participants) | 8 | 18 | 15
microU/ml | 6 (2) | 19 (10) | 11 (5)

3. Primary Outcome: Glucose
Time Frame: Baseline to post 8-10days after VLCD
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lean Baseline | Obese Baseline | Obese Post-diet
Number analyzed (Participants) | 8 | 18 | 15
mg/dL | 82 (6) | 87 (9) | 81 (7)

4. Primary Outcome: Leptin
Time Frame: Baseline to post 8-10days after VLCD
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Lean Baseline | Obese Baseline | Obese Post-diet
Number analyzed (Participants) | 8 | 18 | 15
ng/ml | 13 (5) | 43 (12) | 34 (15)

5. Primary Outcome: Acyl Ghrelin
Time Frame: Baseline to post 8-10days after VLCD
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Lean Baseline | Obese Baseline | Obese Post-diet
Number analyzed (Participants) | 8 | 18 | 15
pg/ml | 235 (104) | 78 (55) | 59 (36)

6. Primary Outcome: Insulin Sensitivity From Oral Glucose Tolerance Test (OGTT_SI)
Description: Insulin Sensitivity from Oral Glucose Tolerance Test was estimated using the minimal model method
Time Frame: Baseline to post 8-10days after VLCD
Population: 9 lean enroll but only 8 complete. A ll lean complete study after baseline outcome measurements.
  19 obese enroll but only 18 complete baseline studies and of these 15 completed the VLCD
Measure: Mean (Standard Deviation); unit: 10-4*min-1*microU-1*mL
Arm/Group | Lean Baseline | Obese Baseline | Obese Post-diet
Number analyzed (Participants) | 8 | 18 | 15
10-4*min-1*microU-1*mL | 11 (4) | 4 (3) | 4 (3)

7. Secondary Outcome: Binge Eating Score Questionnaire
Description: Increased scores indicate increased binge eating behaviors. Score 0-46
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score from questionnaire
Arm/Group | Lean | Obese
Number analyzed (Participants) | 8 | 18
score from questionnaire | 6 (6) | 12 (7)

ADVERSE EVENTS:
Arm/Group | Lean | Obese
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/19
Other Adverse Events (participants affected / at risk) | 0/9 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes